CLINICAL TRIAL: NCT04619823
Title: Virological and Immunological Determinants of Arbovirus Infection in New Caledonia
Acronym: VIRIMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Institut Pasteur de Nouvelle-Calédonie (Unknown); Centre Hospitalier Territorial de Nouvelle-Calédonie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-062
Record Dates: First submitted 2020-09-18; First posted 2020-11-06 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Arbovirus Infections; Zika; Dengue; Chikungunya
Keywords: New Caledonia
MeSH Terms: conditions — Arbovirus Infections; Zika Virus Infection; Dengue; Chikungunya Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient infected by arboviruses (Other)
  Interventions: Other: Blood sample collection

INTERVENTIONS:
Other: Blood sample collection — Blood sample collection Mosquito collection at home

SUMMARY:
Arboviruses, diseases transmitted to humans by the bite of an insect vector, are a major public health problem, particularly in tropical and sub-tropical countries. In New Caledonia, dengue epidemics are recurrent and may be associated with the co-circulation of other arboviruses such as Zika or chikungunya.

The virological determinants which condition the occurrence of these epidemics may be linked to an increased vectorial competence of the vector mosquito Aedes aegypti for a particular viral isolate. In fact, the Aedes aegypti mosquito is infected by making a blood meal on a person infected with an arbovirus. The virus infects its digestive tract, then spreads throughout the mosquito's body until it reaches its salivary glands. The virus is then present in the saliva and will be injected into the human host during a new blood meal. Some viral variants are best transmitted by Aedes aegypti. In general, the study of this vectorial competence is carried out by experiments in the laboratory during which an artificial blood meal composed of mammalian blood (human, rabbit, etc.) is mixed with a viral stock. Carrying out deported blood meals during which blood collected from patients infected with an arbovirus is used to gorge mosquitoes makes it possible to place oneself in experimental conditions as close as possible to the natural cycle of transmission of arboviruses.

In the human host, cells of the myeloid lineage present in the peripheral blood constitute preferred targets of replication for arboviruses. At the same time, the peripheral blood cells of patients are activated in response to infection and secrete many soluble factors released into the blood of patients. The study of blood samples from patients infected with arboviruses is therefore of prime importance for understanding both the replicative mechanisms of arboviruses but also the immune response they induce.

DETAILED DESCRIPTION:
Collection of blood samples from adult patients with clinical signs suggestive of arbovirus

This study is a interventional study that present minimal risks and constraints.

This study will improve :

* the reliability of the results of vector competence experiments
* the understanding of the mechanisms of infection and replication of arboviruses
* the knowledge of the immune mechanisms involved in the response to infection by an arbovirus

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient with clinical signs suggestive of an arbovirus infection:

Fever And at least 2 clinical signs suggestive of arbovirus among which myalgia, retro-orbital pain, drop in platelets (if data available), digestive symptoms, etc.

* Appearance of clinical signs suggestive of an arbovirus infection in the 7 days preceding the blood sample.
* Patient informed of the performance of the research, the collection of data and biological samples
* Patient who has given their consent to participate in the research by authorizing the collection of data, the collection of an additional blood sample and the use of this sample

Exclusion Criteria:

* Patient suffering from another identified virosis, an inflammatory disease or taking anti-inflammatory drugs
* Pregnant patient
* Patient returning from a trip within 15 days before the onset of the signs,
* Patient for whom the blood sample is incomplete or could not be performed
* Patient's condition, which, in the doctor's opinion, is incompatible with the additional sample required by the study
* Patient not having consented to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Measurement of vector competence parameters of Aedes aegypti (carriers or not of Wolbachia) for arboviruses by vector competence experiments using deported blood meals. | 5 years
  Rate of infection of Aedes aegypti (carriers or not of Wolbachia) for arboviruses
Measurement of vector competence parameters of Aedes aegypti (carriers or not of Wolbachia) for arboviruses by vector competence experiments using deported blood meals. | 5 years
  Measurement of dissemination of Aedes aegypti (carriers or not of Wolbachia) for arboviruses
Measurement of vector competence parameters of Aedes aegypti (carriers or not of Wolbachia) for arboviruses by vector competence experiments using deported blood meals. | 5 years
  Measurement of transmission of Aedes aegypti (carriers or not of Wolbachia) for arboviruses

SECONDARY OUTCOMES:
Molecular characterization of arborviruses strains included in the blood of patients and which may be diffused by mosquitoes carrying Wolbachia or not during deported blood meals | 5 years
  Whole genome sequencing and bioinformatics techniques as well as by in vitro infections of arbovirus strains included in the blood of patients and which may be diffused by mosquitoes carrying Wolbachia or not during deported blood meals
Molecular characterization of arborviruses strains contained in mosquitoes present in patients' homes | 5 years
  Whole genome sequencing and bioinformatics techniques as well as by in vitro infections of arbovirus strains contained in mosquitoes present in patients' homes

CONTACTS AND LOCATIONS:
Overall Officials: Myrielle Dupont-Rouzeyrol, PhD, Principal Investigator — Institut Pasteur de Nouvelle-Calédonie
Locations (1):
- Centre Hospitalier Territorial de Nouvelle-Calédonie, Dumbéa Sur Mer, New Caledonia